CLINICAL TRIAL: NCT01709994
Title: Effect of Aspirin in Primary Prevention of Cardiovascular Risk in Patients With Chronic Kidney Disease (AASER Study)
Brief Title: Primary Cardiovascular Risk Prevention With Aspirin in Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación de Ayuda a la Investigación sobre la Hipertensión, Riesgo Cardiovascular y Enfermedades Renales (Other)
Responsible Party: Principal Investigator, Jose Luño Fernandez, Headmaster of Nephrology Department, Fundación de Ayuda a la Investigación sobre la Hipertensión, Riesgo Cardiovascular y Enfermedades Renales
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MG001
Record Dates: First submitted 2012-10-17; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 3
Keywords: cardiovascular events; chronic kidney disease; bleedings; progression; antiinflammatory effects
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aspirin (Active Comparator): Aspirin dosage 100 mg/day
  Interventions: Drug: Aspirin
- standard medication (No Intervention): the patients will continue with standard medication

INTERVENTIONS:
Drug: Aspirin — 100 mg/day of aspirin
  Other Names: ACETILSALYCILIC ACID
  Arms: aspirin

SUMMARY:
The objective of the study is to examine whether the use of low-dose aspirin (75-100 mg / day) reduces the risk of cardiovascular disease in patients with chronic kidney disease (stage 3 or 4).

DETAILED DESCRIPTION:
Hypothesis: The low-dose aspirin reduces cardiovascular risk in patients with chronic kidney disease without increasing the risk of bleeding

ELIGIBILITY:
Inclusion Criteria:

* sign informed consent
* males 45-79 years or females 55-79 years. -Stage 3 or 4 CKD (estimated GFR by MDRD abbreviated, between 15 and 60 ml / min/1.73 m2) -

Exclusion Criteria:

* a previous cardiovascular event: cardiac arrhythmias, cardiac arrest, angina or acute myocardial infarction, stroke, carotid stenosis of more than 50%, peripheral vascular arteriopathy documented
* hospitalization for any cause in the last three months prior to inclusion in the study allergy of acetyl-salicylic acid
* coagulopathy from any cause
* thrombocytopenia <150,000 platelets
* liver disease from any cause
* Infection by hepatitis B virus, hepatitis C or HIV
* immunosuppressive treatment within 12 weeks before inclusion in the study
* Major bleeding events including gastrointestinal bleeding and brain hemorrhage.
* hemoglobinopathies (eg sickle cell disease or thalassemia of any kind)
* active malignancy (except non-melanoma skin cancer). May be included in the study patients with malignant neoplasia who have remained disease-free for at least the previous 5 years.
* uncontrolled inflammatory disease or symptomatic (eg rheumatoid arthritis, lupus, Chrom disease or bowel inflammatory disease)
* hemolysis
* treatment with oral anticoagulation and / or antiplatelet therapy prior.
* poorly controlled hypertension (> 160/90 mm Hg) -pregnancy or breast-
* women of childbearing potential not using effective contraception.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | five years
  To assess the benefit of treatment with low-dose aspirin in the primary prevention of cardiovascular events (incidence of the composite endpoint: death, acute coronary syndrome, stroke or nonfatal acute peripheral arteriopathy disease) in patients with chronic kidney disease who are not in dialysis or renal transplant.

SECONDARY OUTCOMES:
Major bleeding | five years
  -Evaluate the incidence of major bleeding requiring hospitalization
antiinflammatory effects of aspirin | five years
  -to analyze the antiinflammatory effect of aspirin in patients with chronic kidney disease

OTHER OUTCOMES:
progression of chronic kidney disease | five years
  to Analyze the progression of CKD

CONTACTS AND LOCATIONS:
Overall Officials: JOSE LUÑO, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Goicoechea M, de Vinuesa SG, Quiroga B, Verde E, Bernis C, Morales E, Fernandez-Juarez G, de Sequera P, Verdalles U, Delgado R, Torres A, Arroyo D, Abad S, Ortiz A, Luno J. Aspirin for Primary Prevention of Cardiovascular Disease and Renal Disease Progression in Chronic Kidney Disease Patients: a Multicenter Randomized Clinical Trial (AASER Study). Cardiovasc Drugs Ther. 2018 Jun;32(3):255-263. doi: 10.1007/s10557-018-6802-1. PMID 29943364